CLINICAL TRIAL: NCT06059261
Title: A Prospective, Single-arm, Phase II Study of Envafolimab Combined With Chemoradiotherapy and Recombinant Human Endostatin in Locally Advanced Nasopharyngeal Carcinoma.
Brief Title: Envafolimab Combined With Chemoradiotherapy and Recombinant Human Endostatin for LA-NPC.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Collaborators: Fujian Cancer Hospital (Other Government); Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, JiangDong Sui, Deputy Director of Chongqing University Cancer Hospital, Chongqing University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lance
Record Dates: First submitted 2023-09-23; First posted 2023-09-28 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — envafolimab; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab and recombinant human endostatin combined with chemoradiotherapy (Experimental): Intervention Description: Induction envafolimab combined with recombinant endostatin and gemcitabine and cisplatin therapy for three cycles (every 3 weeks) followed by definitive radiotherapy with concurrent cisplatin chemotherapy. After 4 weeks of the completion of radiotherapy, adjuvant envafolimab therapy will begin every 3 weeks for 8 cycles or continue until progression or unacceptable toxicity.
  Interventions: Drug: Envafolimab and recombinant human endostatin combined with chemoradiotherapy

INTERVENTIONS:
Drug: Envafolimab and recombinant human endostatin combined with chemoradiotherapy — Induction treatment phase: Envafolimab administered by subcutaneous injection on day 1 every 3 weeks at 300 mg for 3 cycles, cisplatin administered by intravenous infusion on day 1 of each cycle at 80 mg/m2 every 3 weeks for 3 cycles, gemcitabine was administered by intravenous infusion on days 1 and 8 of each cycle at 1 g/m2 every 3 weeks for 3 cycles, recombinant human endostatin was administered on day 1 every 3 weeks at 210 mg for 3 cycles. Concurrent treatment phase: Cisplatin was administered by intravenous infusion on day 1 of each cycle at 100mg/m2 every 3 weeks for 2 cycles. Adjuvant treatment Phase: Envafolimab was administered on day 1 every 3 weeks at 300 mg for 8 cycles as a subcutaneous injection. Intensity-modulated radiotherapy: 69.96Gy/33fractions/7 weeks,5 fractions/week, 1 fraction/day.

SUMMARY:
This is a multicenter, prospective, single-arm, phase II clinical study, to evaluate the therapeutic efficacy and safety of envafolimab combined with chemoradiotherapy and recombinant human endostatin in patients with locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This is a multicenter, prospective, single-arm phase II clinical study. Patients with high-risk locally advanced stage III-IVA (8th AJCC/UICC staging) primary nasopharyngeal carcinoma, i.e., T4N+ or N2-3, or pretreatment EBV-DNA ≥4000 copies/ml, or lymph node extra-envelope invasion grade 3 (invasion of muscle skin, etc.) are enrolled. After being screened to meet the enrolment criteria and signing the informed consent form, they will receive 3 cycles of induction therapy with envafolimab combined with recombinant human vascular endothelial inhibitor and gemcitabine and cisplatin, followed by cisplatin-concomitant radiotherapy, and 8 cycles of adjuvant therapy with envafolimab after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG score 0-1.
2. Aged 18-65 years, male or non-pregnant female;
3. Pathologically confirmed diagnosis of nasopharyngeal non-keratinizing carcinoma (differentiated or undifferentiated, WHO type II or III) without the need to detect MSI and dMMR status.
4. high-risk locally advanced stage III-IVA (8th AJCC/UICC staging), i.e., T4N+ or N2-3, or pretreatment EBV-DNA ≥4000 copies/ml, or lymph node extra-envelope invasion grade 3 (invasion of muscle skin, etc.), treatment-naive nasopharyngeal carcinoma patients.
5. MRI data of nasopharynx and neck before enrollment, and measurable lesions;
6. Agree to provide a previously stored tumor tissue specimen or biopsy to collect tumor lesion tissue and send it to the central laboratory for PD-L1 IHC testing.
7. Agree to undergo EBV antibody and EBV-DNA quantitative testing before receiving treatment.
8. Hematology: WBC ≥ 4000/μL, neutrophils ≥ 2.000/μL, hemoglobin ≥ 9 g/dL, platelets ≥ 100,000/μL;
9. Liver function: ALT, AST < 1.5 times the upper limit of normal (ULN), total bilirubin < 1.5 × ULN;
10. Renal function: serum creatinine < 1.5 × ULN.
11. Patients have signed the informed consent form and are willing and able to comply with the study plan visits, treatment plan, laboratory tests and other study procedures;

Exclusion Criteria:

1. Patients with recurrent nasopharyngeal carcinoma and distant metastasis.
2. Pathology was keratinizing squamous cell carcinoma (WHO classification type I).
3. Patients who have undergone radiotherapy or systemic chemotherapy;
4. Pregnant or lactating women, in the reproductive period without effective contraceptive measures;
5. HIV positive.
6. Having had other malignancies (except cured basal cell carcinoma or cervical carcinoma in situ);
7. Patients who have been treated with inhibitors of immune regulatory points (CTLA-4, PD-1, PD-L1, etc.);
8. Patients need long-term use of immunosuppressive drug therapy, or systemic or local use of immunosuppressive doses of corticosteroids complications;
9. Patients with immunodeficiency disease, history of organ transplantation (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism; patients with vitiligo or complete remission of asthma in childhood, without any intervention after adulthood can be included; patients with asthma requiring bronchodilators for medical intervention can not be included;
10. Use of excessive doses of glucocorticoids within 4 weeks.
11. Laboratory test values within 7 days before enrollment do not meet the relevant criteria;
12. Patients with significantly low heart, liver, lung, kidney and bone marrow function.
13. Any other diseases or conditions are contraindications to recombinant human vascular endothelial inhibitors, chemoradiotherapy, immunotherapy (such as active phase of infection, within 6 months after myocardial infarction, symptomatic heart disease including unstable angina pectoris, congestive heart failure or uncontrolled arrhythmia, immunosuppressive therapy);
14. Any arterial thrombosis, embolism or ischemia within 6 months before inclusion for treatment, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack;
15. Severe, uncontrolled medical illness and infection.
16. Concurrent use of other investigational drugs or ongoing other clinical trials;
17. Refusing or unable to sign the informed consent form to participate in the trial.
18. Personality or mental disorders, no civil capacity or limited civil capacity;
19. Hepatitis B surface antigen (HBsAg) positive and peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) ≥ 1000cps/ml.
20. Patients who tested positive for HCV antibody were included in the study only if they tested negative for HCV RNA by polymerase chain reaction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-04 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | 3 years
  Defined as the time interval from randomization to tumor progression or death due to any cause. The appearance of new lesions was used as a criterion for progression, and the landmark time point of progression was the date when measurable new lesions were first observed.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  Overall survival is measured from randomization until death due to any cause or the latest known date alive.
Recurrence-free survival(RFS) | 3 years
  Defined as the time from randomization to documented disease recurrence (distant metastasis or local disease recurrence) or death from any cause, whichever occurs first.
Locoregional Relapse-Free Survival (LRFS) | 3 years
  Defined as the time interval from randomization to the first occurrence of recurrence, or to the last follow-up time if there was no recurrence.
Distant metastases-Free survival (DMFS) | 3 years
  Defined as the time interval from randomization to the occurrence of distant metastasis after treatment, or the time to the last follow-up or death due to other causes if there was no distant metastasis.
Incidence rate of adverse events (AEs) | 3 years
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs, according to the Common Terminology Criteria for Adverse Events, version 5.0.
Compliance | 3 years
  Refers to patients taking the drug according to the prescribed dose and course of treatment, as well as the degree of compliance with the study protocol during the implementation by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang D Sui, Ph.D, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Chen YP, Chan ATC, Le QT, Blanchard P, Sun Y, Ma J. Nasopharyngeal carcinoma. Lancet. 2019 Jul 6;394(10192):64-80. doi: 10.1016/S0140-6736(19)30956-0. Epub 2019 Jun 6. PMID 31178151
- [Background] Zhang L, Huang Y, Hong S, Yang Y, Yu G, Jia J, Peng P, Wu X, Lin Q, Xi X, Peng J, Xu M, Chen D, Lu X, Wang R, Cao X, Chen X, Lin Z, Xiong J, Lin Q, Xie C, Li Z, Pan J, Li J, Wu S, Lian Y, Yang Q, Zhao C. Gemcitabine plus cisplatin versus fluorouracil plus cisplatin in recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2016 Oct 15;388(10054):1883-1892. doi: 10.1016/S0140-6736(16)31388-5. Epub 2016 Aug 23. PMID 27567279
- [Background] Mao YP, Xie FY, Liu LZ, Sun Y, Li L, Tang LL, Liao XB, Xu HY, Chen L, Lai SZ, Lin AH, Liu MZ, Ma J. Re-evaluation of 6th edition of AJCC staging system for nasopharyngeal carcinoma and proposed improvement based on magnetic resonance imaging. Int J Radiat Oncol Biol Phys. 2009 Apr 1;73(5):1326-34. doi: 10.1016/j.ijrobp.2008.07.062. Epub 2009 Jan 17. PMID 19153016
- [Background] Li XY, Chen QY, Sun XS, Liu SL, Yan JJ, Guo SS, Liu LT, Xie HJ, Tang QN, Liang YJ, Wen YF, Guo L, Mo HY, Chen MY, Sun Y, Ma J, Tang LQ, Mai HQ. Ten-year outcomes of survival and toxicity for a phase III randomised trial of concurrent chemoradiotherapy versus radiotherapy alone in stage II nasopharyngeal carcinoma. Eur J Cancer. 2019 Mar;110:24-31. doi: 10.1016/j.ejca.2018.10.020. Epub 2019 Feb 7. PMID 30739837
- [Background] Au KH, Ngan RKC, Ng AWY, Poon DMC, Ng WT, Yuen KT, Lee VHF, Tung SY, Chan ATC, Sze HCK, Cheng ACK, Lee AWM, Kwong DLW, Tam AHP. Treatment outcomes of nasopharyngeal carcinoma in modern era after intensity modulated radiotherapy (IMRT) in Hong Kong: A report of 3328 patients (HKNPCSG 1301 study). Oral Oncol. 2018 Feb;77:16-21. doi: 10.1016/j.oraloncology.2017.12.004. Epub 2017 Dec 12. PMID 29362121
- [Background] Sun X, Su S, Chen C, Han F, Zhao C, Xiao W, Deng X, Huang S, Lin C, Lu T. Long-term outcomes of intensity-modulated radiotherapy for 868 patients with nasopharyngeal carcinoma: an analysis of survival and treatment toxicities. Radiother Oncol. 2014 Mar;110(3):398-403. doi: 10.1016/j.radonc.2013.10.020. Epub 2013 Nov 11. PMID 24231245
- [Background] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Adjuvant chemotherapy in patients with locoregionally advanced nasopharyngeal carcinoma: Long-term results of a phase 3 multicentre randomised controlled trial. Eur J Cancer. 2017 Apr;75:150-158. doi: 10.1016/j.ejca.2017.01.002. Epub 2017 Feb 22. PMID 28235726
- [Background] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591
- [Background] Peng H, Chen L, Zhang J, Li WF, Mao YP, Zhang Y, Liu LZ, Tian L, Lin AH, Sun Y, Ma J. Induction Chemotherapy Improved Long-term Outcomes of Patients with Locoregionally Advanced Nasopharyngeal Carcinoma: A Propensity Matched Analysis of 5-year Survival Outcomes in the Era of Intensity-modulated Radiotherapy. J Cancer. 2017 Feb 10;8(3):371-377. doi: 10.7150/jca.16732. eCollection 2017. PMID 28261337
- [Background] Hui EP, Ma BB, Leung SF, King AD, Mo F, Kam MK, Yu BK, Chiu SK, Kwan WH, Ho R, Chan I, Ahuja AT, Zee BC, Chan AT. Randomized phase II trial of concurrent cisplatin-radiotherapy with or without neoadjuvant docetaxel and cisplatin in advanced nasopharyngeal carcinoma. J Clin Oncol. 2009 Jan 10;27(2):242-9. doi: 10.1200/JCO.2008.18.1545. Epub 2008 Dec 8. PMID 19064973
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Jiang XD, Dai P, Wu J, Song DA, Yu JM. Inhibitory effect of radiotherapy combined with weekly recombinant human endostatin on the human pulmonary adenocarcinoma A549 xenografts in nude mice. Lung Cancer. 2011 May;72(2):165-71. doi: 10.1016/j.lungcan.2010.09.003. Epub 2010 Oct 20. PMID 20965604
- [Background] Jain RK. Normalization of tumor vasculature: an emerging concept in antiangiogenic therapy. Science. 2005 Jan 7;307(5706):58-62. doi: 10.1126/science.1104819. PMID 15637262
- [Background] Guan Y, Li A, Xiao W, Liu S, Chen B, Lu T, Zhao C, Han F. The efficacy and safety of Endostar combined with chemoradiotherapy for patients with advanced, locally recurrent nasopharyngeal carcinoma. Oncotarget. 2015 Oct 20;6(32):33926-34. doi: 10.18632/oncotarget.5271. PMID 26418895